CLINICAL TRIAL: NCT02736526
Title: Long-term Prospective Randomized Controlled Clinical Study on Surgical Treatment of Moderate Intermittent Exotropia
Brief Title: Study of Surgical Treatment Versus Observation in Children With Moderate Intermittent Exotropia
Acronym: SOMIX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Tao Shen, M. D., Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZX201304
Record Dates: First submitted 2016-04-03; First posted 2016-04-13 (Estimated); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Moderate Intermittent Exotropia
Keywords: moderate intermittent exotropia; surgical treatment; observation

ARMS (2):
- Surgical treatment (Experimental): The recession or resection of the horizontal extraocular muscles will be processed in the beginning of the trial.
  Interventions: Procedure: recession or resection of the horizontal extraocular muscles
- Observation only (No Intervention)

INTERVENTIONS:
Procedure: recession or resection of the horizontal extraocular muscles
  Arms: Surgical treatment

SUMMARY:
The purpose of this study is to determine the long-term effect and security of the surgical treatment and observation only on ocular alignment, binocular stereopsis, and quality of life in children with moderate intermittent exotropia.

ELIGIBILITY:
Inclusion Criteria:

1. To correspond the definition of IXT: monocular or binocular alternative exotropia, exodeviation at distance for 15 prism diopters at least, can control the normal ocular alignment, normal ocular movements.
2. Simultaneous perception and fusion point in synoptophore, but no normal function of fusion and stereopsis.
3. Age at from 5 to 18 years, sex unlimited.
4. No treatment for IXT previously (including surgical and non-surgical treatment).
5. No amblyopia.
6. Signed informed consent form voluntarily.

Exclusion Criteria:

1. Accompanied with ocular organic diseases.
2. Accompanied with systemic diseases (e.g. nervous system disease).
3. Unable to regular follow-up (e.g. from countryside and outlying district).
4. Investigators concluded that should be excluded.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 280 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Ocular alignment (Prism alternative cover test) | 5 years
Binocular stereopsis at distance and near (Random dot stereopsis test) | 5 years

SECONDARY OUTCOMES:
Newcastle control scores | 5 years
The intermittent exotropia questionnaire | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Shen T, Chen J, Kang Y, Deng D, Lin X, Wu H, Li J, Wang Z, Qiu X, Jin L, Yan J. Surgical treatment versus observation in moderate intermittent exotropia (SOMIX): study protocol for a randomized controlled trial. Trials. 2023 Mar 1;24(1):153. doi: 10.1186/s13063-023-07189-0. PMID 36855155